CLINICAL TRIAL: NCT06322576
Title: A Phase 2, Single-Arm, Multi-center Study of 177Lu-PSMA (177Lu-PNT2002) in Patients With PSMA-Positive Adenoid Cystic Carcinoma
Brief Title: 177Lu-PSMA (177Lu-PNT2002) in PSMA-Positive Adenoid Cystic Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor is no longer producing the study drug, so it was not possible to complete the study.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Adenoid Cystic Carcinoma Research Foundation (Other); Progenics Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00347750
Record Dates: First submitted 2024-02-13; First posted 2024-03-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Adenoid Cystic Carcinoma
Keywords: Lutetium-177
MeSH Terms: conditions — Carcinoma, Adenoid Cystic

STUDY DESIGN:
Intervention Model Description: Cohort 1of this study involves only Dosimetry for (10 patients).
  (Cohort 2 may be added based on dosimetry analysis of Cohort 1. Planned Treatment for would be for 20 patients, single arm).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SPECT CT Dosimetry (Experimental): Absorbed dose in tumor and normal organs will by measured using SPECT/CT dosimetry in Cohort 1.
  Interventions: Drug: 177Lu-PNT2002

INTERVENTIONS:
Drug: 177Lu-PNT2002 — 10 patients will undergo DCFPyL PET/CT and 177Lu-PSMA dosimetry imaging only (single tracer dose).
  If opened, Cohort 2 patients will receive 4 cycles, every 8 weeks of 177Lu-PSMA infusion. Other procedures during treatment and follow up may include: physical exam, CT/MRI, PSMA-PET, blood draws, adverse event assessment, and completion of questionnaires.
  Other Names: 177Lu PSMA

SUMMARY:
This is a single arm trial with one Cohort for people with recurrent or metastatic adenoid cystic carcinoma that cannot be treated with surgery. 10 participants will be enrolled in Cohort 1 at Johns Hopkins and will undergo DCFPyL PET/CT and 177Lu-PSMA dosimetry imaging only (single tracer dose). A feasibility analysis of dosimetry will be performed after meeting the accrual goal of Cohort 1 to determine if the study will proceed into Cohort 2.

If Cohort 2 proceeds, based on the dosimetry analysis, the major requirements of the study are to undergo treatment with 177Lu-PNT2002, have bloodwork, physical exams, and imaging done at study-specific time points, and to answer questionnaires. Patients will be in the study for about two years after enrolling.

DETAILED DESCRIPTION:
Malignant salivary gland tumors account for approximately 3% to 5% of all head and neck cancers with approximately 0.4 to 2.6 cases per 100,000 people. Most patients present in the sixth to seventh decade of life. Adenoid cystic carcinoma (ACC) accounts for about 10% of all tumors of the salivary glands, often arises from the minor and major salivary glands but can also involve lacrimal and ceruminous glands, as well as other sites in the head and neck (nasal and paranasal sinuses, trachea, and larynx). Anatomically, ACC originates from the intercalated duct region and proliferates in three distinct architectural patterns: tubular, cribriform, and solid.

In the setting of recurrent and metastatic (R/M) ACC, first-line options include single-agent vinorelbine or mitoxantrone, or cyclophosphamide plus doxorubicin plus cisplatin (CAP). Overall response rates (ORR) are usually less than 15%. There are no effective second line options. While epidermal growth factor receptor (EGFR) has been shown to be overexpressed in some ACC, none of the phase II clinical trials of single agent cetuximab, gefitinib, or lapatinib demonstrated an objective response. Many cases of ACC also express the c-kit protein, however, use of single agent imatinib in patients with c-kit expression confirmed by immunohistochemistry (IHC) failed to produce an objective response. Phase II single agent sunitinib exhibited no objective response. Median progression free survival (PFS) of these phase II trials ranged from 3.5 months to 7.2 months. Ultimately, most patients with R/M ACC die from cancer, highlighting the need for effective therapies.

The investigators aim to examine and analyze PSMA-PET uptake in ACC to establish whether it is correlated to absorbed tumor dose and objective response in Cohort 1 participants.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation of ACC (primary or metastatic tumor). Central review not required but local pathology review required (at Johns Hopkins or Stanford).
* Patients must have recurrent or metastatic ACC with measurable disease per RECIST 1.1, not amenable to definitive surgery or radiotherapy.
* Patients must have at least 1 lesion positive on PSMA-PET, as defined by standard uptake value (SUV) ratio of tumor to liver greater than one.
* Patient can have any or no prior systemic therapies.
* At least 28 days must have elapsed between last anti-cancer treatment administration and the initiation of study treatment, or at least 5 half-lives of the prior systemic therapy must have elapsed (whichever is shorter).
* Patient must have resolution of all previous treatment related toxicities to CTCAE version 5.0 grade of ≤ 2.
* Patient must be ≥ 18 years of age.
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.

For female patients with childbearing potential or male patients with partners of childbearing potential, agreement to use barrier contraceptive method (condom) and to continue its use for 6 months from receiving the last dose of 177Lu-PSMA. Female patients with childbearing potential will undergo a urine pregnancy test. Pregnant female participants are excluded.

* Patient must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Spinal cord compression or impending spinal cord compression.
* Suspected pulmonary and/or liver metastases (greater >10 mm in largest axis).
* Unable to lie flat during or tolerate PET/CT.
* Refusal to sign informed consent.
* Any medical comorbidities that might preclude safe participation in the study.

Additional inclusion criteria only relevant if Cohort 2 participants enrolled:

* Adequate bone marrow reserve and organ function as demonstrated by complete blood count and chemistry panel completed within the prior 28 days demonstrating:

  1. Platelet count of >100 x109/L
  2. White blood cell (WBC) count > 3,000/mL
  3. Neutrophil count of > 1,500/mL
  4. Hemoglobin ≥ 10 g/dL
  5. Estimated glomerular filtration rate (eGFR) > 50 mL/min based upon Chronic Kidney Disease- Epidemiology Collaboration (CKD-EPI) equation. Due to safety concerns relating to renal clearance and toxicity of 177Lu-PSMA, patients with estimated GFR between 50 - 60 mL/min will require a 99mTc-TPA GFR test and only patients with non-obstructive pathology will be included in the study.
  6. Aspartate transaminase (AST) and alanine aminotransferase (ALT) ≤5 x upper limit of normal (ULN), total bilirubin < 3 x ULN
  7. Total bilirubin < 3 x ULN (except if confirmed history of Gilbert's disease)
  8. Serum albumin > 30 g/L

Additional exclusion criteria only relevant if Cohort 2 participants enrolled:

* Inadequate bone marrow reserve and organ function as detailed in eligibility criteria.
* Patient is participating in a concurrent investigative treatment protocol involving radiotherapy, surgery, or systemic anti-cancer agents.
* Patient receiving any other investigational agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-11-16 (Actual); Study Completion 2026-01-20 (Actual)

PRIMARY OUTCOMES:
Absorbed dose in tumor and normal organs | One dose during one day
  Objective is to measure absorbed dose in tumor and normal organs using SPECT/CT dosimetry (Cohort 1)
Objective response rate (ORR) by RECIST 1.1 measured in patients treated with 177Lu-PSMA for recurrent and metastatic ACC. | Pre-treatment, 6 months post treatment
  Only relevant for Cohort 2 patients: Measure response rate (ORR) by RECIST 1.1 in participants treated with 177Lu-PSMA for recurrent and metastatic ACC.

SECONDARY OUTCOMES:
Stability of Disease: Proportion of patients with Stable Disease | 6 months post treatment
  Cohort 2 participants only. Stability of disease at 6 months is defined as the proportion of patients with SD as assessed per RECIST 1.1 at 6 months after the last cycle of treatment. This 6-month post treatment time point will vary based on the total number of cycles the patient receives.
Progression Free Survival | 24 months after Day 1, Cycle 1 of treatment (each cycle is 8 weeks)
  Only relevant if able to enroll Cohort 2 patients: The distribution of progression free survival will be plotted using the Kaplan Meier method and median values will be estimated and reported with 95% CIs
Overall Survival | 24 months after Day 1, Cycle 1 of treatment (each cycle is 8 weeks)
  Only relevant if able to enroll Cohort 2 patients: The distribution of overall survival will be plotted using the Kaplan Meier method and median values will be estimated and reported with 95% CIs
Duration of Response | 24 months after Day 1 of treatment
  Cohort 2 participants only. Objective response will be defined as evidence of CR, PR, or stable disease. The duration of response will be measured from the start of treatment until the criteria for progression are met.
  Duration of CR or PR: The duration of response (DoR) of CR or PR will be recorded from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that current or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
  Duration of Stable Disease: Stable disease is measured from the start of the treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since the treatment started.
Xerostomia questionnaire (XQ) score | 24 months after Day 1 of treatment
  Only relevant if able to enroll Cohort 2 patients: Xerostomia questionnaire (XQ) will be completed by patients at baseline, prior to each dose of 177Lu-PSMA, at end of treatment, and at follow up visits. XQ measures severity of radiation-induced xerostomia and patient reported quality of life. 8 question total:4 on dryness while eating/chewing, 4 on dryness when not eating/chewing. 0-10 (higher scores=severe dryness/discomfort). Composite Scores range from 0 (no xerostomia) -100 (highest level of xerostomia).
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Head and Neck Module (EORTC QLQ-HN43) | 24 months after Day 1 of treatment
  Only relevant if able to enroll Cohort 2 patients: European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Head and Neck Module (EORTC QLQ-HN43) will be completed by patients at baseline, prior to each dose of 177Lu-PSMA, at end of treatment, and at follow up visits. Answers given according to a 4-point Likert scale, and then transformed so that 0% indicated least symptoms, and 100% most symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Kiess, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Seifert R, Kessel K, Schlack K, Weckesser M, Bogemann M, Rahbar K. Radioligand therapy using [177Lu]Lu-PSMA-617 in mCRPC: a pre-VISION single-center analysis. Eur J Nucl Med Mol Imaging. 2020 Aug;47(9):2106-2112. doi: 10.1007/s00259-020-04703-3. Epub 2020 Feb 16. PMID 32062682
- [Background] von Eyben FE, Roviello G, Kiljunen T, Uprimny C, Virgolini I, Kairemo K, Joensuu T. Third-line treatment and 177Lu-PSMA radioligand therapy of metastatic castration-resistant prostate cancer: a systematic review. Eur J Nucl Med Mol Imaging. 2018 Mar;45(3):496-508. doi: 10.1007/s00259-017-3895-x. Epub 2017 Dec 16. PMID 29247284
- [Background] Rahbar K, Schmidt M, Heinzel A, Eppard E, Bode A, Yordanova A, Claesener M, Ahmadzadehfar H. Response and Tolerability of a Single Dose of 177Lu-PSMA-617 in Patients with Metastatic Castration-Resistant Prostate Cancer: A Multicenter Retrospective Analysis. J Nucl Med. 2016 Sep;57(9):1334-8. doi: 10.2967/jnumed.116.173757. Epub 2016 Apr 7. PMID 27056618
- [Background] van Boxtel W, Lutje S, van Engen-van Grunsven ICH, Verhaegh GW, Schalken JA, Jonker MA, Nagarajah J, Gotthardt M, van Herpen CML. 68Ga-PSMA-HBED-CC PET/CT imaging for adenoid cystic carcinoma and salivary duct carcinoma: a phase 2 imaging study. Theranostics. 2020 Jan 12;10(5):2273-2283. doi: 10.7150/thno.38501. eCollection 2020. PMID 32089741